CLINICAL TRIAL: NCT03808636
Title: Innovative Reagents for Improving Rapid Diagnosis of Mycobacterial Infections
Acronym: TIKA_TB
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: St George's, University of London (Other)
Responsible Party: Sponsor
Other Study IDs: 15.0046
Record Dates: First submitted 2016-01-11; First posted 2019-01-17 (Actual); Last update posted 2019-01-17 (Actual); Status verified 2019-01

CONDITIONS: Tuberculosis (TB)
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TB patients: Any patient with possible or diagnosed tuberculosis who is capable to give informed consent will be offered to be included in the trial

SUMMARY:
The purpose of this study is to quantitate the speed of new culture method using 'Tika' media and compare with conventional systems

DETAILED DESCRIPTION:
Introduction M. tuberculosis (TB) is a significant public health problem in the United Kingdom and abroad. A total of 7832 cases were reported in the UK in 2013. Of those that were culture confirmed (59%) the rate of drug resistance was 7.8%. In certain populations the incidence of drug resistance is higher: homeless patients, those who have been in prison and particularly those from Eastern Europe. Typically the patient will be on treatment for 18 months or more and the PHE has estimated the cost of this as being upto £50000.

Current diagnosis rests on the culture of the M. tuberculosis and drug sensitivity testing. This can take six or eight weeks, meaning that patients may be on ineffective therapy for some time, leading to further transmission and deterioration of the patient's clinical condition. If the speed of culture of the organism could be increased substantially then the delays in diagnosis and getting the correct treatment started could be reduced. In addition if the percentage of culture confirmed cases could be increased then the patient and clinician would benefit. Often patients are started on TB treatment without a confident culture confirmed diagnosis. Other mycobacteria may masquerade as TB causing delays in diagnosis and treatment uncertainty before the confirmed culture result becomes available.

Tuberculosis will be diagnosed in the usual way, by routine analysis of appropriate samples, including standard PCR and culture. Patients who are thought to have or have been confirmed to have tuberculosis will be recruited to the trial.

The patients will be managed in the usual way according to the standard protocols for treating tuberculosis as directed by the treating physician.

Currently the diagnosis of tuberculosis is a lengthy process requiring several weeks of culture of the organism. Identification of a quicker or easier test that might be performed on samples would have great benefits to future patients. The investigators of this research are looking to see if this different method of culture will significantly increase the speed of diagnosis.

Primary Aim To quantitate the speed of new culture method and compare with conventional systems.

This is an observational study and no additional interventions will be performed.

Methods

At least 200 sputum samples obtained from eligible enrolled patients in duplicate:

1. Routine Sample will be labelled and processed by the local NHS Trust Medical Microbiology Department using conventional methods and validated SOP's, as usual.
2. Test sample will be link anonymised and processed as quickly as practical in a separate Category III research laboratory at SGUL by trained research staff.This will extract mycobacteria from the sample which will then be inoculated into a novel media supplemented with growth additives (TiKa Medium). Each Test Sample will then be randomly allocated to one of three different commercially available culture bottle systems (MGIT, BacTAlert, VersaTrek) and processed as usually recommended by the manufacturer for up to 42 days. Time to positivity (TTP) will be recorded and the identity of the growing culture verified using conventional (molecular probe) methodology.

TTP values will be collated in a database. At the end of the study this database will be compared with retrospective data from routine mycobacterial culture results determined from the original parallel samples.

Data analysis will determine the degree of improvement (as determined in days to positivity) delivered by each method and will test the hypothesis that the TiKa Medium can significantly (P<0.05) improve the recovery of non-culturable phenotypes and make culturable phenotypes of pathogenic mycobacteria grow faster from clinical samples, than previously observed.

There will be no exceptions (waivers) to eligibility criteria prior to participant inclusion into the study. Any questions raised about eligibility should be addressed prior to entering the participant.

Inclusion criteria: Any patient with possible or diagnosed tuberculosis who is capable to give informed consent will be offered to be included in the trial.

Exclusion criteria: Any patient under 18 or who is unable to give informed consent will be excluded from this trial. Any persons under detention will not be included. Any patient who is unable to give a sample.

Any patient may withdraw from the study at any time. Any patients who are lost to follow up will be contacted and attempts will be made to re-engage them with services as is standard practice for patients with tuberculosis.

Participant recruitment at a site will only commence once evidence of the following approval/essential documents are in place:

1. The main REC approval, if applicable
2. Final sponsorship and host site approval,

All participants who wish to enter the study will be fully screened and consented by the Chief Investigator, or one of the qualified clinicians involved in the study as Clinical Co-investigator.

Patients will be approached by the routine clinical team and asked if they would be interested. If they express an interest one of the researchers will contact them.

Consent will be taken by a member of the research team who has had experience, training and qualifications in Good Clinical Practice around taking consent.

A copy of the signed Informed Consent Form (ICF) along with a copy of the Patient Information Sheet (PIS) will be given to the study participant. An original signed & dated consent form will be retained in the medical notes and a copy will be placed in the ISF.

At enrollment data will be collected in pseudoanonymised form as per protocol.

All data will be handled in accordance with the Data Protection Act 1998. The Case Report Forms (CRFs) will not bear the participant's name or other directly identifiable data. The participant's trial Identification Number (ID) only, will be used for identification. The sponsor Subject ID log JREOLOG0002 can be used to cross reference participant's identifiable information.

Case Report Forms will be designed by the CI and the final version will be approved by the Sponsor. All data will be entered legibly in black ink with a ball-point pen as per GCP.

The agreed archiving period for this trial will be 5 years. This will include any study databases.

The number of patients to be enrolled in the study has been calculated using a standard power calculation based upon previous experimental data suggesting that an effect size of >0.3 would be achievable within the standard deviation expected using this protocol at an error probability of 0.05. This would estimate a 0.95 power to be 20% below the number of sample expected to collect.

Primary endpoint: To show statistical difference (P<0.05) between Test and Routine group sample TTP data.

Statistical analysis plan: Summary of baseline data and flow of patients. The researchers are proposing to enroll 200 patients over a period of 9 months. The research site is a centre of excellence and referral for tuberculosis and the researchers fully expect to meet this participant number. There is no differential patient treatment involved in this study and there will be no requirement to randomise patients within the study.

Test samples however will be randomised post processing for inclusion in each of the three culture machines (arms) using a random number generated chart (n=3) limited to provide equal numbers to each test arm.

This study is fully financed with funding from Innovate UK

ELIGIBILITY:
Inclusion Criteria:

* Any patient with possible or diagnosed tuberculosis who is capable to give informed consent will be offered to be included in the trial.

Exclusion Criteria:

* Any patient under 18 or who is unable to give informed consent will be excluded from this trial.
* Any persons under detention will not be included. Any patient who is unable to give a sample.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient with possible or diagnosed tuberculosis
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2015-06; Primary Completion 2019-03 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Time of culture growth using the new culture method | one year
  To quantitate the speed of new culture method systems.

SECONDARY OUTCOMES:
Difference between the times of new and conventional culture methods. | one year
  Comparison of the speed of the new culture method with conventional systems.

CONTACTS AND LOCATIONS:
Overall Officials: Tim Bull, PhD, Study Director — St George's Univeristy of London; Catherine Cosgrove, PhD MRCP, Principal Investigator — St George's Univeristy of London
Locations (1):
- St George's NHS Healthcare Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Samples are anonymised

REFERENCES:
- See also: Number and proportion of culture confirmed cases by country, PHE 2013 — https://www.gov.uk/government/uploads/system/uploads/attachment_data/file/358254/TB_culture_confirmed_cases_by_country_and_PHE_centre__2013_.pdf